CLINICAL TRIAL: NCT05313867
Title: Effects of Dietary Supplements Based on Trace Elements on Voice Parameters and Some Psychological and Physiological Parameters Related to Stress - Single-center, Comparative, Cross-over, Randomized, Double-blind Study Versus Placebo, in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Pronutri (Industry)
Collaborators: Clin-Experts (Industry); Plateforme Cocolab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2021-A02571-40
Record Dates: First submitted 2022-03-20; First posted 2022-04-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Stress
Keywords: Stress; trace elements; voice parameters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1 sequence of 10 tablets containing only excipients
  Interventions: Dietary Supplement: Placebo
- Trace elements (Experimental): Nutri VX1 in a single dose (1 sequence of 10 tablets). Nutri VX1 is a complex of trace elements with the status of a food supplement.
  Interventions: Dietary Supplement: Nutri VX 1

INTERVENTIONS:
Dietary Supplement: Nutri VX 1 — 1 sequence of 10 tablets (one intake)
  Arms: Trace elements
Dietary Supplement: Placebo — 1 sequence of 10 tablets (one intake)
  Arms: Placebo

SUMMARY:
Preliminary data obtained by the company Pronutri, which produces food supplements based on trace metals, suggests that food supplements containing trace metal compounds could act by reducing stress, which could result in effects on various physiological parameters.

Trace elements are pure minerals essential to the functioning of our body, present in very small quantities. They have a precise and fundamental role in biological and information processes: a deficiency can lead to dysfunctions, often at the origin of our daily ailments.

No scientific study has so far been carried out to measure the effects of these molecules on physiological and psychological parameters related to stress in healthy volunteers. The present study therefore aims to test the effects of these tablets containing metals and trace metals on the reduction of stress.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Healthy (healthy volunteers) (no current treatment except contraception and no acute illness within 3 months)
* Affiliated to the social security system
* Signed consent

Exclusion Criteria:

* Voice disorders: aphasia, dysphonia, aphonia...
* Presence of a cardiac pacemaker
* Person intolerant to lactose, or to any excipient present in the VX 1 product
* Person under legal protection or unable to give consent
* Minor
* Pregnant or post-pregnant woman under 6 months or of childbearing age without effective contraception
* Person deprived of liberty by a judicial or administrative decision or under psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
F0 voice frequency | Change from baseline at 5 minutes after the intake
  The vocal parameters will be evaluated using the Praat software (duration of sound in sec, average duration of pauses in sec, average vocal frequency expressed in Hz (F0), standard deviation of F0 expressed in Hz, minimum and maximum of F0, "jitter " and "shimmer"

CONTACTS AND LOCATIONS:
Overall Officials: Alice GUYON, Principal Investigator — Plateforme Cocolab - Maison des Sciences de l'Homme et de la Société Sud-Est
Locations (1):
- Plateforme Cocolab - Maison des Sciences de l'Homme et de la Société Sud-Est, 24, avenue des Diables Bleus, Campus Saint Jean d'Angély, Nice, France

IPD SHARING:
Plan to Share IPD: No